CLINICAL TRIAL: NCT00864968
Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Nabumetone 750 mg Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-493
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Nabumetone; Healthy subjects
MeSH Terms: interventions — Nabumetone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Nabumetone 750 mg tablets, single dose
  Interventions: Drug: Nabumetone 750 mg tablets, single dose
- B (Active Comparator): Nabumetone 750 mg tablets, single dose
  Interventions: Drug: Nabumetone 750 mg tablets, single dose

INTERVENTIONS:
Drug: Nabumetone 750 mg tablets, single dose — A: Experimental Subjects received Actavis Elizabeth LLC formulated products under fasting conditions
  Other Names: Nabumetone
  Arms: A
Drug: Nabumetone 750 mg tablets, single dose — B: Active comparator Subjects received Teva formulated products under fasting conditions
  Other Names: Nabumetone
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of nabumetone from 2 tablet products and determine if the 2 products were bioequivalent to each other.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Nabumetone 750 mg Tablets in Healthy Volunteers

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria

1. Healthy subjects at least 18 years of age.
2. Availability of the subject for the entire study period and willingness to provide written informed consent after being informed of the nature of the study.
3. Body mass index (BMI) between 18 and 30 kg/m2 (calculated using the BMI Calculator on the Centers for Disease Control and Prevention [CDC] website available at http://www.cdc.gov/nccdphp/dnpa/bmi/index.htm, last accessed 19 Mar 07) and a weight of at least 110 pounds.
4. Good health as determined by a lack of clinically significant abnormalities in health assessments performed at Screening, as judged by the physician.
5. Females were required to use a medically acceptable method of hormonal contraception or abstinence throughout the entire study period and for one week after the study is completed

Exclusion Criteria

1. Hypersensitivity to nabumetone (Nabumetone) or related compounds.
2. Conditions that affected the absorption, metabolism, or passage of drugs out of the body (eg, sprue, celiac disease, Crohn's disease, colitis, liver, kidney, or thyroid conditions).
3. Recent history (within 1 year) of mental illness, drug addiction, drug abuse, or alcoholism.
4. A hematocrit value of ≤ 33.0% for females and ≤ 37.0% for males.
5. Donation of > 500 mL of blood in the past 8 weeks prior to study drug dosing or difficulty in donating blood.
6. Receipt of an investigational drug within the 4 weeks prior to study drug dosing.
7. Currently taking any systemic prescription medications, excluding hormone contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition did not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications, as judged by the attending physician.

   Any nonprescription medication consumption reported was to be reviewed by the investigator prior to dosing. At the discretion of the investigator, these volunteers could be enrolled if the medication was not anticipated to alter study integrity.
8. Regular smoking of more than 5 cigarettes weekly or the regular daily use of nicotinecontaining products beginning 3 months before study drug administration through the final evaluation.
9. Female subjects who were lactating or had a positive pregnancy test at Screening and prior to each of the treatment periods.
10. Alcohol, grapefruit beverages or foods, caffeine, or xanthine beverages or foods beginning 48 hours before each study drug administration through the last pharmacokinetic (PK) sample of each treatment period. Such restricted items included coffee, tea, iced tea, Coke®, Pepsi®, Mountain Dew®, chocolate, brownies, etc.
11. Regular use of any drugs known to induce or inhibit hepatic drug metabolism (examples include barbiturates, carbamazepine, rifampin, phenylhydantoins, phenothiazines, cimetidine, omeprazole, macrolides, imidazoles, fluoroquinolones) within 30 days prior to study drug administration.
12. Positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C antibody at Screening.
13. Positive test results for drugs of abuse or pregnancy at Screening and prior to each study drug dosing period. Any deviation from these inclusion and exclusion criteria must have been approved by the investigator and/or the sponsor on a case-by-case basis prior to enrollment of the subject. The protocol deviation waiver must have been documented by the investigator and/or the sponsor.

No subject was allowed to enroll in this study more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Evin H. Sides III, M.D., Principal Investigator — AAIPharma Inc., AAI Clinic
Locations (1):
- AAIPharma Inc., AAI Clinic, Morrisville, North Carolina, United States